CLINICAL TRIAL: NCT02706418
Title: A Standardised Massage Protocol as an Effective Treatment for Chronic Carpal Tunnel Syndrome
Brief Title: Clinical Massage Therapy as a Treatment for Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jing Advanced Massage Training (Other)
Collaborators: Medway NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTS-01
Record Dates: First submitted 2016-02-26; First posted 2016-03-11 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

ARMS (1):
- Clinical Massage Therapy (Other)
  Interventions: Procedure: Clinical Massage Therapy

INTERVENTIONS:
Procedure: Clinical Massage Therapy

SUMMARY:
Once participants have been recruited, their grip strength shall be tested and they will all complete baseline questionnaires to assess functional status and symptom severity.

Following the recruitment stage, participants will be asked to attend Medway Maritime Hospital once a week for four weeks, to receive the massage protocol. At the first session participants shall be asked to rate their pain (NPRS), before receiving a massage treatment. This will be followed by instructions on how to perform self-massage, which they will be asked to complete daily over the four-week period, and record in a diary. At the remaining three sessions, participants shall just complete the NPRS prior to receiving the massage treatment.

After four weeks the group will be reassessed at the same Orthopaedic Clinic they attended prior to recruitment. They will be asked to complete a final pain score, record any changes in their condition, repeat the initial symptom questionnaire, and finally preform a grip strength test. The duration of four weeks was chosen as this is the time-frame within which the specific massage protocol advises a 'significant symptom improvement' should be seen.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or above.
* Pain paraesthesia and/or hypoesthesia in the hand, in the area innervated by the median nerve.
* Participants must have a clinical diagnosis of Carpal Tunnel Syndrome (CTS).
* Participant must be able to comply with the study procedures.
* Participant must have attended the Medway Maritime Hospital (Kent), for assessment of the present condition.
* Participant is willing and able to give informed consent for participation in the study.
* Participant must not be contra-indicated for the receipt of massage.
* Participants must be able to speak and read English fluently.

Exclusion Criteria:

* Participants who are receiving any additional treatment for their carpal tunnel pain that is not part of standard care (topical pain relief, bracing).
* Participants that have had any surgery on the anatomical sites relevant to the condition and/or treatment (neck, shoulder, arm, wrist, hand).
* Participants that have any suggestion of an additional condition related to carpal tunnel pain (i.e. previous trauma, pregnancy, etc).
* Planning to undertake any activities or lifestyle changes which may affect their levels of carpal tunnel pain (e.g. changing/ceasing occupation, alternative symptom therapy, adopting/ceasing a hobby).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Number of participants experiencing improvements in the symptoms of Carpal Tunnel Syndrome as assessed by the Boston Carpal Tunnel Questionnaire (BCTQ), change from baseline in the symptom severity scores at 4 weeks. | 4 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Medway Maritime Hospital, Gillingham, Kent, United Kingdom